CLINICAL TRIAL: NCT00801697
Title: A Phase 1B Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant Adenoviral Subtype 35 (rAd35) and Subtype 5 (rAd5) HIV-1 Vaccines When Given as a Heterologous Prime-boost Regimen or as Boosts to a Recombinant DNA Vaccine in Healthy, Ad5-Naïve and Ad5-Exposed, Low Risk, HIV-1 Uninfected Adult Participants
Brief Title: Safety and Immune Response to Preventive HIV Immunization With Adenovirus Serotype 5 or 35 Vector
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 077; 10702 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine; Adenovirus
MeSH Terms: conditions — HIV Infections; Adenoviridae Infections | interventions — Vaccines, DNA

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (8):
- 1A (Experimental): rAD5-naive participants will receive rAd35 intramuscularly at study entry and rAd5 intramuscularly at Month 6
  Interventions: Biological: rAd35; Biological: rAd5
- 1B (Placebo Comparator): Participants will receive rAd35 placebo intramuscularly at study entry and rAd5 placebo intramuscularly at Month 6
  Interventions: Biological: rAd35 placebo; Biological: rAd5 placebo
- 2A (Experimental): rAD5-naive participants will receive DNA vaccine intramuscularly at study entry and Months 1 and 2 and rAd5 intramuscularly at Month 6
  Interventions: Biological: DNA Vaccine; Biological: rAd5
- 2B (Placebo Comparator): Participants will receive DNA vaccine placebo intramuscularly at study entry and Months 1 and 2 and rAd5 placebo intramuscularly at Month 6
  Interventions: Biological: DNA Vaccine placebo; Biological: rAd5 placebo
- 3A (Experimental): Participants will receive DNA vaccine intramuscularly at study entry and Months 1 and 2 and rAd35 intramuscularly at Month 6
  Interventions: Biological: DNA Vaccine; Biological: rAd35
- 3B (Placebo Comparator): Participants will receive DNA vaccine placebo intramuscularly at study entry and Months 1 and 2 and rAd35 placebo intramuscularly at Month 6
  Interventions: Biological: DNA Vaccine placebo; Biological: rAd35 placebo
- 4A (Experimental): Participants will receive DNA vaccine intramuscularly at study entry and Months 1 and 2 and rAd35 intramuscularly at Month 6
  Interventions: Biological: DNA Vaccine; Biological: rAd35
- 4B (Placebo Comparator): Participants will receive DNA vaccine placebo intramuscularly at study entry and Months 1 and 2 and rAd35 placebo intramuscularly at Month 6
  Interventions: Biological: DNA Vaccine placebo; Biological: rAd35 placebo

INTERVENTIONS:
Biological: DNA Vaccine — 4 mg VRC-HIVDNA044-00-VP administered as 1 mL
  Arms: 2A; 3A; 4A
Biological: DNA Vaccine placebo — 1 mL VRC-PBSPLA043-00-VP
  Arms: 2B; 3B; 4B
Biological: rAd35 — VRC-HIVADV027-00-VP 1 x 10^10 PU administered as 1 mL
  Arms: 1A; 3A; 4A
Biological: rAd35 placebo — 1 mL VRC-PBSPLA043-00-0VP
  Arms: 1B; 3B; 4B
Biological: rAd5 — 4 mg VRC-HIVADV038-00-VP administered as 1 mL
  Arms: 1A; 2A
Biological: rAd5 placebo — 1 mL VRC-DILUENT013-DIL-VP
  Arms: 1B; 2B

SUMMARY:
This study will evaluate the safety and preliminary immune response to recombinant adenoviral serotype 35 and 5 HIV-1 vaccines in HIV-uninfected adults.

DETAILED DESCRIPTION:
One of the more promising approaches in the development of a preventive HIV vaccine uses a DNA plasmid to prime the immune response to an adenoviral vector boost. This primary purpose of this study is to evaluate the safety, tolerability, and immune response to recombinant adenoviral serotype 35 (rAd35) and serotype 5 (rAD5) HIV-1 vaccines in Ad-5 naive and Ad-5 exposed HIV-uninfected adults.

This study will last approximately 12 months. Participants will include those who are both rAD5-naive and rAD5-exposed and will be stratified into one of four groups. Each group will consist of two arms, one interventional and one control. Participants in Groups 1, 2, and 3 will be rAD5-naive. Participants in Group 4 will be rAD5-exposed.

Participants in Group 1 will receive an injection of rAD35 vaccine or placebo at study entry and an injection of rAD5 vaccine or placebo at Month 6 with nine follow-up visits through Month 12. Participants in Groups 2, 3, and 4 will injections of DNA vaccinations or placebo at study entry and at Months 1 and 2, and an injection of rAD35 vaccine, rAD5 vaccine, or placebo at Month 6 with twelve follow-up visits though Month 12. A physical, questionnaire, and counseling will occur at all visits. Blood and urine collection will occur at most visits. A rectal swab will occur at selected visits. For females, a pregnancy test will occur at all visits.

Participants will be contacted for safety follow-ups after the injection every year for 5 years. Health and adverse events will be recorded. Participants will not need to return to the study clinic unless HIV confirmatory testing is needed.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Access to a participating HVTN clinical research site and willingness to be followed for the duration of the study
* Assessment of understanding, including understanding of Step Study results
* Willing to receive HIV test results
* Willing to discuss HIV infection risks, agree to HIV risk reduction counseling, and willing to continue 5 years of annual follow-up contact
* Willing to commit to maintaining behavior consistent with low risk of HIV exposure through the last required protocol visit
* Considered low risk for HIV infection after clinical staff assessment. More information on this criterion can be found in the protocol.
* Certain laboratory values. More information on this criterion can be found in the protocol.
* Negative Hepatitis B surface antigen
* Negative anti-Hepatitis C virus antibodies
* For females, agree to use effective contraception from at least 21 days prior to enrollment through the last protocol visit. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* HIV-infected
* Active drug or alcohol abuse within 12 months prior to study entry
* History of newly acquired sexually transmitted infections. More information on this criterion can be found in the protocol.
* Experimental vaccines received within 5 years prior to study entry
* Immunosuppressive medications received within 168 days prior to first vaccination
* Blood products received within 120 days prior to first vaccination
* Immunoglobulin received within 60 days prior to first vaccination
* Live attenuated vaccines received within 30 days prior to first vaccination
* Investigational research agents received within 30 days prior to first vaccination
* Intent to participate in another study of an investigational research agent during planned duration of the study
* Any vaccines that not live attenuated vaccines and were received within 14 days prior to first vaccination
* Allergy treatment with antigen injections within 30 days prior to first vaccination or scheduled within 14 days after first vaccination
* Clinically significant medical condition, findings, results, or history with implications for current health. More information on this criterion can be found in the protocol.
* Serious adverse reactions to vaccines
* Autoimmune disease
* Immunodeficiency
* Active Syphilis infection within the past 6 months
* Asthma. More information on this criterion can be found in the protocol.
* Diabetes mellitus
* Thyroidectomy or thyroid disease requiring medication during the last 12 months
* Hypertension. More information on this criterion can be found in the protocol.
* Body mass index greater than 35 or 40. More information on this criterion can be found in the protocol.
* Bleeding disorder
* Malignancy
* Seizure disorder
* Asplenia
* Psychiatric condition that precludes compliance with the protocol
* Any other clinically significant condition or laboratory abnormality that, in the opinion of the investigator, would interfere with the study
* Pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Local and systemic reactogenicity signs and symptoms, laboratory measures of safety, and adverse and expedited adverse events | Throughout study
Magnitude and frequency of immune responses between HIV-1 clade A env rAD35 and rAd5 vaccines when given as a boost after DNA vaccine | At Week 4 following the fourth vaccination
Magnitude and frequency of immune responses between clade A env rAD35 vaccine primed by Ad35 versus DNA | At Week 4 following the last vaccination
Magnitude and frequency of immune responses of HIV-1 clade A env rAD35 vaccine when given as a boost | At Week 4 following the fourth vaccination

SECONDARY OUTCOMES:
Immunogenicity of HIV-1 clade A env rAD35 vaccine given as a prime | At Week 4 following the first vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Fuchs, MD, MPH, Study Chair — SFDPH/UCSF; Pierre-Alexandre Bart, MD, Study Chair — CHUV (Lausanne)
Locations (10):
- United States (10):
  - Alabama CRS, Birmingham, Alabama
  - Bridge HIV CRS, San Francisco, California
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Fenway Health (FH) CRS, Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee
  - Seattle Vaccine and Prevention CRS, Seattle, Washington

REFERENCES:
- [Background] Buchbinder SP, Mehrotra DV, Duerr A, Fitzgerald DW, Mogg R, Li D, Gilbert PB, Lama JR, Marmor M, Del Rio C, McElrath MJ, Casimiro DR, Gottesdiener KM, Chodakewitz JA, Corey L, Robertson MN; Step Study Protocol Team. Efficacy assessment of a cell-mediated immunity HIV-1 vaccine (the Step Study): a double-blind, randomised, placebo-controlled, test-of-concept trial. Lancet. 2008 Nov 29;372(9653):1881-1893. doi: 10.1016/S0140-6736(08)61591-3. Epub 2008 Nov 13. PMID 19012954
- [Background] Priddy FH, Brown D, Kublin J, Monahan K, Wright DP, Lalezari J, Santiago S, Marmor M, Lally M, Novak RM, Brown SJ, Kulkarni P, Dubey SA, Kierstead LS, Casimiro DR, Mogg R, DiNubile MJ, Shiver JW, Leavitt RY, Robertson MN, Mehrotra DV, Quirk E; Merck V520-016 Study Group. Safety and immunogenicity of a replication-incompetent adenovirus type 5 HIV-1 clade B gag/pol/nef vaccine in healthy adults. Clin Infect Dis. 2008 Jun 1;46(11):1769-81. doi: 10.1086/587993. PMID 18433307
- [Background] Sheets RL, Stein J, Bailer RT, Koup RA, Andrews C, Nason M, He B, Koo E, Trotter H, Duffy C, Manetz TS, Gomez P. Biodistribution and toxicological safety of adenovirus type 5 and type 35 vectored vaccines against human immunodeficiency virus-1 (HIV-1), Ebola, or Marburg are similar despite differing adenovirus serotype vector, manufacturer's construct, or gene inserts. J Immunotoxicol. 2008 Jul;5(3):315-35. doi: 10.1080/15376510802312464. PMID 18830892
- [Derived] Fischinger S, Cizmeci D, Deng D, Grant SP, Frahm N, McElrath J, Fuchs J, Bart PA, Pantaleo G, Keefer M, O Hahn W, Rouphael N, Churchyard G, Moodie Z, Donastorg Y, Streeck H, Alter G. Sequence and vector shapes vaccine induced antibody effector functions in HIV vaccine trials. PLoS Pathog. 2021 Nov 29;17(11):e1010016. doi: 10.1371/journal.ppat.1010016. eCollection 2021 Nov. PMID 34843602